CLINICAL TRIAL: NCT03831555
Title: Use of a Psychosocial Readiness Tool to Improve Hepatitis C Treatment Adherence and Outcomes at the Grady Liver Clinic
Brief Title: Tool to Improve Treatment Adherence and Outcomes at Grady Liver Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lesley Miller, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00093687
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C
Keywords: Psychosocial Readiness Evaluation and Preparation for Hepatitis C Treatment tool
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREP-C (Active Comparator): The research assistant will complete the abbreviated PREP-C survey with the study participants either before or after their medical appointment. The PREP-C tool is accessed online at https://prepc.org/.
  Interventions: Behavioral: PREP-C
- Standard of care (No Intervention): Participants will receive the standard of care (usual care) for chronic HCV infection.

INTERVENTIONS:
Behavioral: PREP-C — The Psychosocial Readiness Evaluation and Preparation for Hepatitis C Treatment (PREP-C) tool assesses a patient's psychosocial readiness to start HCV treatment. There are nine sections in the survey:
  1. Motivation: reasons client wants to begin HCV treatment, concerns about treatment, and the importance of treatment
  2. Information: knowledge about HCV treatment and one's own HCV disease status
  3. Medication Adherence: current prescribed medications and adherence to them in the prior month
  4. Self-efficacy: self-confidence about adhering to HCV treatment
  5. Social Support and Stability: stability of financial, housing, and social support resources
  6. Alcohol and substance use: alcohol and substance use behaviors and current treatment
  7. Psychiatric Stability: current psychiatric status, previous and current treatment
  8. Energy Level: sleep and fatigue
  9. Cognitive Functioning: perceived difficulty with communication in health care setting, problem-solving ability, and memory.
  Arms: PREP-C

SUMMARY:
The purpose of this study is to learn more about what psychological and social factors affect people in how they take their hepatitis C medications.

DETAILED DESCRIPTION:
The goal of this study is to determine if a qualitative survey that assesses a patient's readiness for treatment of Hepatitis C (HCV) and associated interventions based on identified barriers can improve treatment adherence and outcomes. HCV remains a leading cause of liver cancer and end stage liver disease despite greater than 90% cure rates with new, all-oral antiviral medications. While these new medications are easier to tolerate and access than previous treatment regimens, medication adherence still remains a great barrier to cure. In this study, we will administer the Psychosocial Readiness Evaluation and Preparation for Hepatitis C Treatment (PREP-C) tool, a free, online survey developed at the Mount Sinai School of Medicine to determine psychosocial readiness for treatment.

ELIGIBILITY:
Inclusion Criteria:

* seen in the Grady Liver Clinic during the study time period
* have a confirmed chronic hepatitis C infection (hepatitis C antibody positive and detectable hepatitis C viral load)

Exclusion Criteria:

* no chronic hepatitis C infection
* co-infection with HIV or hepatitis B
* non-English speaking
* unable to consent to participate
* already started HCV therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants keeping follow-up appointments | At 4 months
  Adherence to HCV treatment will be measured by documenting the number of participants keeping their follow-up appointments. This data will be collected from chart reviews.
Number of participants keeping follow-up appointments | At 8 months
  Adherence to HCV treatment will be measured by documenting the number of participants keeping their follow-up appointments. This data will be collected from chart reviews.
Number of participants refilling medications | At 4 months
  Adherence to HCV treatment will be measured by documenting the number of participants who refill their medications. This data will be collected from chart reviews.
Number of participants refilling medications | At 8 months
  Adherence to HCV treatment will be measured by documenting the number of participants who refill their medications. This data will be collected from chart reviews.
Number of participants who keep lab visits | At 4 months
  Adherence to HCV treatment will be measured by documenting the number of participants who keep their lab visits.This data will be collected from chart reviews.
Number of participants who keep lab visits | At 8 months
  Adherence to HCV treatment will be measured by documenting the number of participants who keep their lab visits.This data will be collected from chart reviews.
Rapid virologic response (RVR) | At 4 weeks
  The treatment outcome will be measured by analyzing the rapid virologic response (RVR) at 4 weeks after completion of treatment. Rapid virologic response (RVR) is defined as an undetectable serum hepatitis C virus (HCV) RNA. This data will be collected from chart reviews.
Sustained virologic response (SVR) | At 12 weeks
  The treatment outcome will be measured by analyzing the sustained virologic response (SVR) at 12 weeks after completion of treatment. SVR is defined as aviremia 12 weeks after completion of antiviral therapy. This data will be collected from chart reviews.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Miller, MD, Principal Investigator — Emory University
Locations (1):
- Grady Liver Clinic, Atlanta, Georgia, United States